CLINICAL TRIAL: NCT05578599
Title: A Prospective, Single-center Clinical Pilot Study Evaluating Feasibility of the Swiftsure Complete Care System (CCS) in Intubated Adults Undergoing Mechanical Ventilation
Brief Title: A Pilot Study Swiftsure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22-554
Record Dates: First submitted 2022-09-28; First posted 2022-10-13 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Ventilated Patients

STUDY DESIGN:
Intervention Model Description: Single arm study - treatment with the Swiftsure CSS device in addition to standard oral care procedures. Using a measuring scale of 1 to 5, for each patient, whereas 1 is low outcome of standard oral care and using the Swiftcare device, and 5 is best results for using standard oral care and the Swiftcare device.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental Treatment (Other): Treatment with the Swiftsure CSS device in addition to standard oral care procedures
  Interventions: Device: Swiftsure CCS device

INTERVENTIONS:
Device: Swiftsure CCS device — The Swiftsure CSS device will be used twice per patient in addition to standard oral health care procedures among intubated adult patients undergoing mechanical ventilation in the ICU.

SUMMARY:
The purpose of this study is to investigate the feasibility of using the Swiftsure Complete Care System (CCS) device as an adjunct to standard oral care procedures among intubated adult patients undergoing mechanical ventilation in the intensive care unit (ICU).

This is a small study intended to gather initial feasibility before conducting a larger study. The feasibility of using the Swiftsure CSS device will be studied among 20 patients at a single study site.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, non-blinded trial to assess the feasibility of using the Swiftsure CSS device as an adjunct to the standard oral care among intubated adult patients undergoing mechanical ventilation in the ICU.

The CSS intervention will be performed 1 times per subject. The nurse performing the intervention will be asked to complete the study questionnaires after each device use.

ELIGIBILITY:
Inclusion Criteria:

* Cardio-Vascular Intensive Care Unit (CVICU) patients recovering from surgery and expected to undergo mechanical ventilation for at least 6 hours
* 18 years or older

Exclusion Criteria:

* Unable to consent
* Maxillofacial trauma
* Agitation
* Tested positive for COVID-19 at screening
* Any condition precluding positioning required for device use (e.g. increased intracranial pressure, spine instability, presence of spine drain etc)
* Oropharyngeal injury or infection
* Respiratory infection
* Difficult Airway Grade III or higher
* Intubated with a double lumen tube
* Tracheostomy
* Endotracheal tube cuff air leak, defined as inspiratory-to-expiratory tidal volume difference higher than 10% or audible gurgling at cuff pressure higher than 30 cmH2O
* Poor dental status
* Hemodynamic instability, defined as need for 2 or more vasopressor agents, or use of mechanical hemodynamic support (e.g. intra-aortic balloon pump, Impella heart pump, Left Ventricular Assist Device, venous- arterial extracorporeal membrane oxygenation)
* Respiratory instability, defined as PaO2/FIO2 < 300 mmHg on PEEP > 10 cmH2O, or respiratory acidosis with pHa < 7.30 and respiratory rate > 20, or use of inhaled pulmonary vasodilators
* Pregnancy or not using anti-conceptional agents in child bearing age
* Patients with difficult intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Procedural success | 1 to 4 hours post-procedure
  Procedural success, defined as successful completion of the full procedure to use the Swiftsure CCS device, and standard oral care,

SECONDARY OUTCOMES:
Usability of Swiftsure CCS device | 1 to 4 hours post-procedure
  The investigators will define success as an average score of neutral (i.e. 3) 1 is less or less success and 5 is best sucess, on a 5-point scale as measured by the Device Use Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Gama de Abreu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida VFA, Reuter Pimenta A, Lara-Erazo V, Karki D, Rodriguez-Patarroyo F, Semeia J, Duncan H, Filipovic N, Meyer D, Gama de Abreu M. Swiftsure complete care system in intubated adults: a feasibility study. Expert Rev Med Devices. 2025 Nov;22(11):1265-1270. doi: 10.1080/17434440.2025.2576586. Epub 2025 Oct 24. PMID 41123953